CLINICAL TRIAL: NCT02892266
Title: Prevalence and Correlates of Post-Traumatic Stress Symptoms (PTSS) in Adolescent Solid Organ Transplant Recipients (CTOTC-11)
Brief Title: Post-Traumatic Stress Symptoms (PTSS) in Transplant Recipients
Acronym: CTOTC-11
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Clinical Trials in Organ Transplantation in Children (Other)
Responsible Party: Sponsor
Other Study IDs: DAIT CTOTC-11
Record Dates: First submitted 2016-08-11; First posted 2016-09-08 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Solid Organ Transplant Recipients; Parent(s)/Guardian of Referenced Transplant Recipients
Keywords: Transplant recipients; Adolescents; Post-Traumatic Stress Symptoms (PTSS); Transplant Recipient and Family Impact(s)
MeSH Terms: interventions — Mental Health; Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Adolescent Transplant Recipients: 1. Questionnaire battery at enrollment (Participants and their parents/guardians)
  2. Clinical data from patient's chart (6 months of retrospective data & 6 months of prospective tacrolimus trough level data)
  Interventions: Other: Assessment of adherence, mental health, behavioral, quality of life and biological constructs

INTERVENTIONS:
Other: Assessment of adherence, mental health, behavioral, quality of life and biological constructs

SUMMARY:
This study is conducted to better understand Post-Traumatic Stress Symptoms (PTSS) in adolescent transplant recipients and their parent/guardian and to see if PTSS play a role in the way adolescent transplant recipients take their prescribed medicine.

Target population: medically stable adolescent solid organ (e.g., heart, kidney, liver, lung, small bowel) transplant recipients and their parent(s)/guardian.

ELIGIBILITY:
Inclusion Criteria:

The patient:

* and/or their parent(s)/guardian must be able to understand and provide informed consent in English or Spanish;
* is prescribed tacrolimus (either brand or generic formulation); and
* has been seen in the enrolling center's clinic at least twice in the last two years.

Exclusion Criteria:

The patient:

* received a transplant less than 18 months prior to enrollment;
* has had more than one transplant (including marrow replacement);
* or their parent(s)/guardian is actively psychotic or severely disoriented due to any cause, including hepatic encephalopathy (temporary exclusion);
* or their parent(s)/guardian has been diagnosed with severe intellectual disability as defined in the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5);
* is not medically stable or is hospitalized;
* is currently enrolled in a study that aims to improve adherence to medical recommendations;
* is receiving cognitive behavioral therapy for confirmed or suspected diagnosis of Post-Traumatic Stress Disorder (PTSD) at enrollment;
* is receiving psychotropic medications for a confirmed or suspected diagnosis of PTSD.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Adolescent transplant recipients at risk for non-adherence and can reliably answer self-report questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2016-09; Primary Completion 2018-11-24 (Actual); Study Completion 2018-11-24 (Actual)

PRIMARY OUTCOMES:
Medication Level Variability Index (MLVI) | 6 months retrospective data to 6 months post enrollment
  Defined by fluctuation in medication blood levels. Calculated as the standard deviation (variation) of a minimum of 3 outpatient tacrolimus trough levels, obtained for one year, consisting of 6 months prior to study enrollment plus 6 months post study enrollment.
University of California at Los Angeles Post-Traumatic Stress Disorder Reaction Index DSM-5 (UCLA PTSD RI DSM-5) Total Score | At enrollment visit
  The UCLA PTSD RI DSM-5 is a widely used and validated self-report questionnaire assessing posttraumatic stress symptoms (PTSS) in children and adolescents ages 8-18 years.

SECONDARY OUTCOMES:
Above-threshold Medication Level Variability Index (MLVI) | 6 months post enrollment
  Defined by an MLVI greater than 2.
Above-threshold Child PTSS Score | At enrollment visit
  Defined as the existence of threshold scores in a symptoms constellation corresponding to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) definition of Post-Traumatic Stress Disorder (PTSD). Method: University of California at Los Angeles Post-Traumatic Stress Disorder Reaction Index DSM-5 version (UCLA PTSD RI DSM-5) self-report questionnaire.
Child Avoidance Score | At enrollment visit
  Measured by the UCLA Post-Traumatic Stress Disorder Reaction Index (PTSD-RI) self-report subscale summary score.
Parent PTSS Total Score | At enrollment visit
  Measured using the Impact of Event Scale (IES) self-report questionnaire.
Parent Avoidance | At enrollment visit
  Measured using IES self-report questionnaire subscore.
Diagnosis of chronic allograft rejection | 6 months retrospective data to 6 months post enrollment
Diagnosis of graft failure | 6 months retrospective data to 6 months post enrollment
Child Depression/Distress Assessment | At enrollment visit
  Depression/distress measured using the Children's Depression Inventory - Short Form (CDI-S) self-report questionnaire.
Quality of Life (QOL) Assessment Using the PedsQL Total Score | At enrollment visit
  Measured using the child self-report Pediatric Quality of Life (PedsQL) version 4.0.
QOL Assessment Using PedsQL Subscale Scores | At enrollment visit
  Measured using the child self-report PedsQL version 4.0 subscale scores.
QOL Assessment Using the HRQOL (PedsQL) Total Score | At enrollment visit
  Measured using the child self-report Transplant-Specific Health-Related Quality of Life (HRQOL) scale (PedsQL) version 4.0 summary score.
PedsQL Family Impact Total Score | At enrollment visit
  Measured using the parent/guardian self-report PedsQL Family Impact version 2.0 summary score.
PedsQL Family Impact Subscale Scores | At enrollment visit
  Measured using the parent/guardian self-report PedsQL Family Impact version 2.0 subscale scores.
Types of traumas identified as salient by the child | At enrollment visit
  Measured using the University of California at Los Angeles Post-Traumatic Stress Disorder Reaction Index DSM-5 version (UCLA PTSD RI DSM-5).
Types of traumas identified as salient by the parent | At enrollment visit
  Measured using the parent/guardian Impact of Event Scale (IES).

OTHER OUTCOMES:
Exploratory Outcome: Dose of steroids | At enrollment
  Potential impact of steroid use on PTSD will be assessed by a correlation coefficient between mean steroid dose per kilogram.
Exploratory Outcome: Presence of Donor Specific Antibodies (DSA) | At enrollment Visit

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Sweet, M.D., Ph.D., Study Chair — St. Louis Children's Hospital: Pediatric Transplantation
Locations (13):
- United States (13):
  - Ronald Reagan UCLA Medical Center: Pediatric Transplantation, Los Angeles, California
  - Lucile Salter Packard Children's Hospital at Stanford: Pediatric Transplantation, Palo Alto, California
  - UCSF Benioff Children's Hospital: Pediatric Transplantation, San Francisco, California
  - University of Miami, Jackson Memorial Hospital: Pediatric Transplantation, Miami, Florida
  - Ann and Robert H. Lurie Children's Hospital of Chicago: Pediatric Transplantation, Chicago, Illinois
  - Boston Children's Hospital: Pediatric Transplantation, Boston, Massachusetts
  - St. Louis Children's Hospital: Pediatric Transplantation, St Louis, Missouri
  - Columbia University Medical Center: Pediatric Transplantation, New York, New York
  - Cincinnati Children's Hospital Medical Center: Pediatric Transplantation, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia: Pediatric Transplantation, Philadelphia, Pennsylvania
  - University of Texas Southwestern/Children's Medical Center: Pediatric Transplantation, Dallas, Texas
  - Texas Children's Hospital: Pediatric Transplantation, Houston, Texas

REFERENCES:
- See also: The National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: The Clinical Trials in Organ Transplantation in Children (CTOT-C) — http://www.ctotc.org/